CLINICAL TRIAL: NCT05665712
Title: Pediatric Enhanced Recovery After Cardiac Surgery: a Single-centre Retrospective Study
Brief Title: Pediatric Enhanced Recovery After Cardiac Surgery
Acronym: PERCS
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00104502
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: ERAS; Pediatric ALL; Congenital Heart Disease
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Heart Defects, Congenital | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: enhanced recovery — bundle of factors that have been shown to help with recovery in other surgical services such as good pain control, early ambulation, early nutrition

SUMMARY:
Identify our institution's current perioperative management strategies for pediatric cardiac surgery patients. Identify predictive factors for receiving perioperative care following P-ERACS strategies.

Compare outcomes between P-ERACS and non-P-ERACS patients

DETAILED DESCRIPTION:
study aims to 1) assess our institution's current perioperative management strategies for pediatric cardiac surgery patients, 2) identify which patient population would be appropriate for inclusion in a pediatric ERACS (P-ERACS) program, and 3) compare the outcomes of patients whose perioperative care followed general consensus P-ERACS strategies (P-ERACS patients) and those whose perioperative care did not (non-P-ERACS patients). Results from this study will inform current efforts to establish a local P-ERACS protocol, and facilitate the initiation of a clinical trial to assess adherence to a P-ERACS pathway as well as the impact of such a pathway on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* all pediatric patients (<18 years of age) who underwent elective cardiac surgery requiring cardiopulmonary bypass (CPB)

Exclusion Criteria:

* Emergency procedures and transplantation (heart, lung, heart and lung)

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: all pediatric patients (<18 years of age) who underwent elective cardiac surgery requiring cardiopulmonary bypass (CPB)
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
time to extubation | 24 hours
  time to extubation

SECONDARY OUTCOMES:
Length of stay | 48 hours
  LOS in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Noss C, Prusinkiewicz C, Nelson G, Patel PA, Augoustides JG, Gregory AJ. Enhanced Recovery for Cardiac Surgery. J Cardiothorac Vasc Anesth. 2018 Dec;32(6):2760-2770. doi: 10.1053/j.jvca.2018.01.045. Epub 2018 Jan 31. PMID 29503121
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Background] Roy N, Parra MF, Brown ML, Sleeper LA, Nathan M, Sefton BA, Baird CW, Mistry KP, Del Nido PJ. Initial experience introducing an enhanced recovery program in congenital cardiac surgery. J Thorac Cardiovasc Surg. 2020 Nov;160(5):1313-1321.e5. doi: 10.1016/j.jtcvs.2019.10.049. Epub 2019 Oct 24. PMID 31859070